CLINICAL TRIAL: NCT02549157
Title: Relationship Between Treatments for Urogynecological Problems and Patient Reported Values, Psychological States, and Quality of Life
Brief Title: Treatments for Urogynaecological Problems and Patient Selfreports
Status: Recruiting | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Principal Investigator, Prof Phil Reed, Professor Phil Reed, Swansea University
Other Study IDs: IRAS project ID: 130775
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Urogynaecological Problem, Pelvic Floor Dysfunction, Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pelvic Floor Muscle Training

SUMMARY:
The research aims to assess the relationship between treatments for a range of urogynaecological problems (pelvic floor dysfunction, cancers) and patient reported values, psychological states, and quality of life. The impact of treatments on patients' health outcomes will be measured, using specific urogynaecological outcome measures (for either pelvic floor dysfunction or cancer), and patient reported measures of general health and quality of life. Patients' psychological states and values will be measured by validated self-report instruments for these areas. Researchers will obtain consent for participation from patients. Following consent, baseline measures will be taken at the patients' routine appointment about 4 weeks prior to undergoing treatment (e.g., surgery or physiotherapy for pelvic floor dysfunction, or surgery for a urogynaecology cancer). These measures will be the routinely collected physical data obtained by medical staff, and patient reported measures of their general health, psychological state, and quality of life. These questionnaires should take about 30 minutes to complete, in total. The patients will undergo treatment (physiotherapy programme or surgery), which will not be affected by this research. About four weeks post treatment, patients will receive their usual appointment, and routinely collected physical data will be obtained by medical staff, and patients will complete the measures as described above. With the patient's consent, the above evaluation will be repeated at every follow-up appointment that the patient has (i.e. after 3months, and then at yearly intervals, for 5 years). The impact of treatments on objective routine health measures taken by medical staff, and on patient reported measures of health, quality of life, personal values, and psychological functioning, will be documented at each measurement point. Additionally, relationships between psychological states/values and both objective and subjective ratings of how treatments have impacted the patients will be established.

DETAILED DESCRIPTION:
Aims The research aims to assess the relationship between treatments for various uro-gynaecological problems (pelvic floor dysfunction, and cancer) and both: (i) objective physical outcomes, and (ii) self reported outcomes in terms of general health, and quality of life, at a number of time points post treatment (4 week, 3months, 1year, and yearly, thereafter).

In addition, the research aims to assess the relationship between psychological factors (depression, anxiety, and values) prior to treatment, and treatment outcomes (specific outcome, self reported general health, and quality of life), at time points post treatment (4 week, 3months, 1year, and yearly, thereafter), for patients with various gynaecological problems (pelvic floor dysfunction, and cancers).

Participants and Recruitment Consecutive patients referred for treatments (physiotherapy, surgery) for uro-gynaecological problems (pelvic floor dysfunction, cancer) will be asked if they would like to participate in this evaluative study. The initial approach will be made through a letter sent out with their appointment details, which will give information about the study. This will make clear that their treatment will not depend on their participation in the study. The patients also will be given the chance to discuss their participation with the specialist nurse at the time of their pre-treatment assessment, and will give their consent (by completing and signing a Consent Form) on the day of their taking part in the research study, after they have had time to think about their participation and ask any questions that they may have.

Design and Methodology Following their consent, at the initial consultation prior to treatment (about 4 weeks prior to treatment), baseline measures will be taken from the patients. These measures will be the routinely collected physical data, obtained by the medical staff, plus a series of patient-reported measures, concerned with the patients' general health (GHQ28), depression and anxiety (HADS), values (PVQII), and quality of life (EQ5D, WHOQoL-BREF, and QLQC30). These questionnaires should take about 30 minutes to complete, in total. The patients will then undergo their treatment (the type of treatment decided upon forms no part of this study). About four weeks post-treatment, the patients will receive their usual physical screening by medical staff, and will, again, complete the same forms as described above. The patients will then be asked if they would complete the same questionnaires at a series of subsequent time points (approximately after 3 months post treatment, and then yearly for five years). The changes across the objectively- and subjectively-reported health status, and in the patient-reported quality of life, and psychological functioning will be measured. Additionally, the relationship between the baseline patient-reported psychological states (depression and anxiety) and values, and the objective (physical measures), and subjectively-reported (general health and quality of life) outcomes, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* consenting patients who are referred for pelvic floor problems to Singleton Hospital Swansea, UK.

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for treatments (physiotherapy, surgery) for urogynaecological problems (pelvic floor dysfunction, cancer) will be asked if they would like to participate in this study. Initial approach will be made through letter sent out with their appointment details, which will give information about the study. This will make clear that their treatment will not depend on their participation in the study. The patients also will be given the chance to discuss their participation with the specialist nurse at the time of their pre-treatment assessment, and will give their consent (by completing and signing a Consent Form) on the day of their taking part in the research study, after they have had time to think about their participation and ask any questions that they may have.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09-01; Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in objective physical outcomes | Initial measures will be taken about 4 weks pre-treatment, and then again 4 weeks post-treatment. Follow-up measures will be taken after abou 3 months, and then after 1 year for each of the next 4 years.
  Oxford Grading
Change in self reported depression and anxiety | Initial measures will be taken about 4 weks pre-treatment, and then again 4 weeks post-treatment. Follow-up measures will be taken after abou 3 months, and then after 1 year for each of the next 4 years.
  Hospital Anxiety and Depresion Scales, ranging from 0-21 for both scales, with 9 or more being considered as showing signs of depression or anxiety.
Change in self reported quality of life | Initial measures will be taken about 4 weks pre-treatment, and then again 4 weeks post-treatment. Follow-up measures will be taken after abou 3 months, and then after 1 year for each of the next 4 years.
  Euro-qual 5D measures health related quality of life on 5 dimensons (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each rated as: "no problems," "slight problems," "moderate problems," "severe problems," and "unable to"/"extreme problems"
Change in personal values | Initial measures will be taken about 4 weks pre-treatment, and then again 4 weeks post-treatment. Follow-up measures will be taken after abou 3 months, and then after 1 year for each of the next 4 years.
  Personal Values Questionnaire measures patient selected areas of their life which they value (e.g., health, family), giving a score between 0 and 25, with higher scores indicating a more strongly heald value.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Reed, D.Phil., Principal Investigator — Swansea University
Locations (1):
- Singleton Hospital, Swansea, United Kingdom

REFERENCES:
- [Derived] Osborne LA, Mair Whittall C, Emery S, Reed P. Change in depression predicts change in bladder symptoms for women with urinary incontinence undergoing pelvic-floor muscle training. Eur J Obstet Gynecol Reprod Biol. 2023 Jan;280:54-59. doi: 10.1016/j.ejogrb.2022.11.010. Epub 2022 Nov 14. PMID 36402023
- [Derived] Reed P, Osborne LA, Whittall CM, Emery S. Impact of patient motivation on compliance and outcomes for incontinence. Physiotherapy. 2021 Dec;113:100-106. doi: 10.1016/j.physio.2020.10.003. Epub 2020 Oct 24. PMID 34563914